CLINICAL TRIAL: NCT02641106
Title: Video Directly Observed Therapy (VDOT) to Monitor Short-Course LTBI Treatment
Brief Title: VDOT for Monitoring Adherence to LTBI Treatment
Acronym: VMALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Richard S Garfein, PhD, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 150155
Record Dates: First submitted 2015-12-20; First posted 2015-12-29 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Tuberculosis; Latent Tuberculosis Infection
Keywords: Telemedicine; Mobile Phone; Adherence; Latent Tuberculosis Infection; Directly Observed Therapy; Video DOT
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis; Directly Observed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Directly Observed Therapy (Experimental): VDOT arm participants use a smartphone to make a video recording of each weekly medication dose ingested using the VDOT mobile phone app. The VDOT app is programmed to send encrypted, time/date stamped videos to a HIPAA-compliant server as soon as the video recorder is stopped. Clinic staff monitor videos as they arrive using a password protected website and document each medication dose that is taken. Dose 1 is observed in-person; doses 2-12 are observed via videos.
  Interventions: Other: Video Directly Observed Therapy
- In-Person DOT (Active Comparator): In-Person DOT arm participants follow standard-of-care procedures for monitoring ingestion of all medication doses. Participants take their first medication dose at the enrollment visit and return to the clinic once weekly to be observed taking the remaining 11 doses of medication until they complete the 12-dose regimen.
  Interventions: Other: In-Person DOT

INTERVENTIONS:
Other: Video Directly Observed Therapy — Video Directly Observed Therapy (VDOT) is a novel means of remotely observing patients ingesting medications using videos sent from a smartphone. VDOT was developed and found to be feasible and acceptable for monitoring daily treatment of active TB in San Diego, CA and Tijuana, B.C., Mexico (R21-AI088326; PI: R. Garfein). Patients are taught how to use the VDOT recording app, record medication ingestion, and contact their physician when side effects occur. Participants are trained at the time of their first LTBI treatment dose to ensure participants know how to record videos. All remaining 11 weekly doses are taken and recorded wherever the participant chooses. Clinic staff monitor videos as they arrive using a password protected website and document each medication dose that is taken.
  Other Names: VDOT
  Arms: Video Directly Observed Therapy
Other: In-Person DOT — Clinic-based, in-person DOT is the standard of care for monitoring adherence for patients taking the 12-dose isoniazid/rifapentine treatment for LTBI. Participants visit the clinic once weekly until all 12 doses are taken or 16 weeks pass, whichever comes first.
  Other Names: Control
  Arms: In-Person DOT

SUMMARY:
The three-month short-course treatment with isoniazid [H] and rifapentine [P] (3HP) recently recommended by the Centers for Disease Control and Prevention could dramatically increase the number of persons starting and completing treatment for latent tuberculosis infection (LTBI), but TB providers nationwide are hamstrung by the requirement that 3HP only be administered by directly observed therapy (DOT) in which patients are watched taking each medication dose in-person. We developed a novel mHealth application that allows patients to make and send videos of each medication dose ingested that are watched by healthcare providers via a HIPAA-compliant website to remotely monitor LTBI treatment adherence (Video DOT [VDOT]). This study will determine whether monitoring patients with VDOT achieves higher treatment completion rates and greater patient acceptability at lower cost than clinic-based in-person DOT.

DETAILED DESCRIPTION:
Building on our novel VDOT System that includes text messaging reminders and HIPAA-compliant cloud-based administration, we hypothesize that VDOT can be expanded to provide higher treatment completion rates at a lower cost than in-person DOT for LTBI treatment using 3HP. We propose a randomized controlled trial to address the following specific aims:

Aim 1: To determine whether LTBI treatment completion and adherence are greater for patients treated with 3HP administered via VDOT versus in-person DOT, and to identify patient factors associated with these outcomes; Aim 2: To compare acceptability of treatment by patients on VDOT versus in-person DOT, and identify factors associated with differences in acceptability; Aim 3: To calculate the cost-effectiveness of VDOT compared to in-person DOT for administering 3HP.

To address the study aims we will conduct a randomized controlled trial in which TB contacts and refugees in San Diego who are prescribed 3HP for LTBI treatment by their physician will be randomly assigned to be monitored for adherence via either VDOT or in-person DOT (Figure 2). Approximately 100 patients per year over three years (n=155/arm) will be recruited through the San Diego County TB Control and Refugee Health Program (TCRHP) clinics for the trial. Patients assigned to VDOT will be given a smartphone with service and taught to send videos of themselves taking each weekly medication dose; patients in the in-person DOT arm will visit the clinic each week to be observed by a healthcare worker taking their LTBI medication. Medication adherence will be monitored for all participants until they have taken all 12 doses or 16 weeks (limit recommended by the CDC to complete treatment), to compare treatment adherence rates and patient acceptance across trial arms. Participants will complete brief (20 minute) baseline and follow-up assessment interviews to obtain information about potential confounders and effect modifiers of adherence and patient acceptance regarding their treatment administration method. Cost-benefit analyses will also be conducted to assist in developing policies around the use of VDOT for 3HP. Since participants will be recruited after they have been prescribed 3HP by their healthcare provider and all patient care will be continued through their provider, no medications will be prescribed or treatment decisions made this study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of LTBI and patient's physician determines that they are eligible to receive 3HP
2. Age ≥13 years;
3. No plans to move out of the San Diego area within 4 months of enrollment; and
4. Willing to comply with study procedures and provide informed consent (or assent for minors and parental consent) prior to study enrollment.

Exclusion Criteria:

1. Are younger than 13 years old;
2. Plan to move out of San Diego County within 4 months of enrollment;
3. Refuse to allow study staff to review their medical records;
4. Are incarcerated;
5. Have a physical (e.g., blindness) or cognitive disabilities that make VDOT impractical unless someone else in their household can assist them for the duration of the study; or
6. Are using other medications that preclude the use of 3HP (e.g., antiretroviral medication for HIV).

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants completing LTBI treatment | 16 weeks
  The proportion of participants completing treatment (i.e., taking all 12 prescribed doses within 16 weeks). At the end of 16 weeks, the participant will have either completed the 12-dose treatment or considered defaulted.
Participant satisfaction with method of monitoring LTBI treatment | 16 weeks
  Compare level of participant satisfaction with treatment by each method of treatment monitoring. After the last dose of medication is taken (or at 16 weeks for those who do not complete treatment), follow-up interviews will collect treatment satisfaction outcome data.
cost-effectiveness of VDOT compared to in-person DOT for administering 3HP | 5 years
  Compare the cost of providing DOT by each method of treatment monitoring. Since this outcome requires program costs for delivery of the VDOT intervention, the time frame for collecting all cost data is 4 years.

SECONDARY OUTCOMES:
Proportion of participants completing LTBI treatment in 12 weeks | 12 weeks
  Proportion of participants completing LTBI treatment on-schedule (i.e., participants took all 12 doses within 12 weeks, as prescribed). By the end of 12 weeks, participants who ingested 12 doses within 12 weeks will be counted as achieving this outcome; all others will be counted failing this outcome.
Proportion of participants who took all 12 LTBI treatment doses on-schedule | 12 weeks
  Proportion of participants completing LTBI treatment on-schedule (i.e., participants took all 12 doses on the same day each week for 12 consecutive, as prescribed). By the end of 12 weeks, participants who ingested 12 doses within 12 weeks on the same day each week will be counted as achieving this outcome; all others will be counted failing this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Garfein, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- San Diego County Health and Human Services Agency, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided